CLINICAL TRIAL: NCT04739800
Title: A Randomized Phase II Trial of Triplet Therapy (A PD-L1 Inhibitor Durvalumab (MEDI4736) in Combination With Olaparib and Cediranib) Compared to Olaparib and Cediranib or Durvalumab (MEDI4736) and Cediranib or Standard of Care Chemotherapy in Women With Platinum-Resistant Recurrent Epithelial Ovarian Cancer, Primary Peritoneal or Fallopian Cancer Who Have Received Prior Bevacizumab
Brief Title: Comparison of Standard of Care Treatment With a Triplet Combination of Targeted Immunotherapeutic Agents
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2021-00615; NCI-2021-00615 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GY023 (Other: NRG Oncology); NRG-GY023 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2021-02-04; First posted 2021-02-05 (Actual); Results first posted 2024-06-18 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-07

CONDITIONS: Fallopian Tube Mucinous Adenocarcinoma; Ovarian Seromucinous Carcinoma; Platinum-Refractory Fallopian Tube Carcinoma; Platinum-Refractory Ovarian Carcinoma; Platinum-Refractory Primary Peritoneal Carcinoma; Recurrent Fallopian Tube Clear Cell Adenocarcinoma; Recurrent Fallopian Tube Endometrioid Adenocarcinoma; Recurrent Fallopian Tube High Grade Serous Adenocarcinoma; Recurrent Fallopian Tube Mucinous Adenocarcinoma; Recurrent Fallopian Tube Transitional Cell Carcinoma; Recurrent Fallopian Tube Undifferentiated Carcinoma; Recurrent Low Grade Fallopian Tube Serous Adenocarcinoma; Recurrent Ovarian Clear Cell Adenocarcinoma; Recurrent Ovarian Endometrioid Adenocarcinoma; Recurrent Ovarian High Grade Serous Adenocarcinoma; Recurrent Ovarian Low Grade Serous Adenocarcinoma; Recurrent Ovarian Mucinous Adenocarcinoma; Recurrent Ovarian Seromucinous Carcinoma; Recurrent Ovarian Transitional Cell Carcinoma; Recurrent Ovarian Undifferentiated Carcinoma; Recurrent Platinum-Resistant Fallopian Tube Carcinoma; Recurrent Platinum-Resistant Ovarian Carcinoma; Recurrent Platinum-Resistant Primary Peritoneal Carcinoma; Recurrent Primary Peritoneal Clear Cell Adenocarcinoma; Recurrent Primary Peritoneal Endometrioid Adenocarcinoma; Recurrent Primary Peritoneal High Grade Serous Adenocarcinoma; Recurrent Primary Peritoneal Low Grade Serous Adenocarcinoma; Recurrent Primary Peritoneal Transitional Cell Carcinoma; Recurrent Primary Peritoneal Undifferentiated Carcinoma; Refractory Fallopian Tube Clear Cell Adenocarcinoma; Refractory Fallopian Tube Endometrioid Adenocarcinoma; Refractory Fallopian Tube High Grade Serous Adenocarcinoma; Refractory Fallopian Tube Mucinous Adenocarcinoma; Refractory Fallopian Tube Transitional Cell Carcinoma; Refractory Fallopian Tube Undifferentiated Carcinoma; Refractory Low Grade Fallopian Tube Serous Adenocarcinoma; Refractory Ovarian Clear Cell Adenocarcinoma; Refractory Ovarian Endometrioid Adenocarcinoma; Refractory Ovarian High Grade Serous Adenocarcinoma; Refractory Ovarian Low Grade Serous Adenocarcinoma; Refractory Ovarian Mucinous Adenocarcinoma; Refractory Ovarian Seromucinous Carcinoma; Refractory Ovarian Transitional Cell Carcinoma; Refractory Ovarian Undifferentiated Carcinoma; Refractory Primary Peritoneal Clear Cell Adenocarcinoma; Refractory Primary Peritoneal Endometrioid Adenocarcinoma; Refractory Primary Peritoneal High Grade Serous Adenocarcinoma; Refractory Primary Peritoneal Low Grade Serous Adenocarcinoma; Refractory Primary Peritoneal Transitional Cell Carcinoma; Refractory Primary Peritoneal Undifferentiated Carcinoma
MeSH Terms: interventions — Specimen Handling; cediranib; Contrast Media; durvalumab; Immunoglobulin G; Disulfides; Magnetic Resonance Spectroscopy; olaparib; Paclitaxel; Taxes; liposomal doxorubicin; Doxorubicin; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm I (paclitaxel, doxorubicin, topotecan hydrochloride)) (Active Comparator): Patients receive paclitaxel IV over 60 minutes on days 1, 8, and 15, or pegylated liposomal doxorubicin hydrochloride IV over 60 minutes on day 1, or topotecan hydrochloride IV over 30 minutes on days 1, 8 and 15 or days 1-5 per the discretion of the treating physician. Cycles repeat every 21 or 28 days in the absence of disease progression or unacceptable toxicity. Patients may undergo ECHO or MUGA during screening and as clinically indicated on study. Patients also undergo collection of blood and CT with contrast during screening, and CT or MRI scans throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Computed Tomography with Contrast; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Drug: Paclitaxel; Drug: Pegylated Liposomal Doxorubicin Hydrochloride; Drug: Topotecan Hydrochloride
- Arm II (durvalumab, cediranib maleate, olaparib) (Experimental): Patients receive durvalumab IV over 60 minutes on day 1, cediranib maleate PO QD Monday through Friday, and olaparib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients may undergo ECHO or MUGA during screening and as clinically indicated on study. Patients also undergo collection of blood and CT with contrast during screening, and CT or MRI scans throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Drug: Cediranib Maleate; Procedure: Computed Tomography; Procedure: Computed Tomography with Contrast; Biological: Durvalumab; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Drug: Olaparib
- Arm III (durvalumab, cediranib maleate) (Experimental): Patients receive durvalumab IV over 60 minutes on day 1 and cediranib maleate PO QD Monday through Friday. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients may undergo ECHO or MUGA during screening and as clinically indicated on study. Patients also undergo collection of blood and CT with contrast during screening, and CT or MRI scans throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Drug: Cediranib Maleate; Procedure: Computed Tomography; Procedure: Computed Tomography with Contrast; Biological: Durvalumab; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan
- Arm IV (cediranib maleate, olaparib) (Experimental): Patients receive cediranib maleate PO QD on days 1-28 and olaparib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients may undergo ECHO or MUGA during screening and as clinically indicated on study. Patients also undergo collection of blood and CT with contrast during screening, and CT or MRI scans throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Drug: Cediranib Maleate; Procedure: Computed Tomography; Procedure: Computed Tomography with Contrast; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Drug: Olaparib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cediranib Maleate — Given PO
  Other Names: AZD2171; AZD2171 Maleate; Recentin
  Arms: Arm II (durvalumab, cediranib maleate, olaparib); Arm III (durvalumab, cediranib maleate); Arm IV (cediranib maleate, olaparib)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Computed Tomography with Contrast — Undergo CT with contrast
  Other Names: Contrast Enhanced Computed Tomography; CONTRAST ENHANCED CT SCAN; Contrast-enhanced Computed Tomography; CT Scan With Contrast; CT with Contrast
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI 4736; MEDI-4736; MEDI4736
  Arms: Arm II (durvalumab, cediranib maleate, olaparib); Arm III (durvalumab, cediranib maleate)
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
  Arms: Arm I (paclitaxel, doxorubicin, topotecan hydrochloride)); Arm II (durvalumab, cediranib maleate, olaparib); Arm III (durvalumab, cediranib maleate)
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU 0059436; KU-0059436; KU0059436; Lynparza; Olanib; Olaparix; PARP Inhibitor AZD2281
  Arms: Arm II (durvalumab, cediranib maleate, olaparib); Arm IV (cediranib maleate, olaparib)
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm I (paclitaxel, doxorubicin, topotecan hydrochloride))
Drug: Pegylated Liposomal Doxorubicin Hydrochloride — Given IV
  Other Names: ATI-0918; Caelyx; Dox-SL; Doxil; Doxilen; Doxorubicin HCl Liposomal; Doxorubicin HCl Liposome; Doxorubicin Hydrochloride Liposome; Duomeisu; Evacet; LipoDox; Lipodox 50; Liposomal Adriamycin; Liposomal Doxorubicin Hydrochloride; Liposomal-Encapsulated Doxorubicin; Pegylated Doxorubicin HCl Liposome; Pegylated Liposomal Doxorubicin; S-Liposomal Doxorubicin; Stealth Liposomal Doxorubicin; TLC D-99
  Arms: Arm I (paclitaxel, doxorubicin, topotecan hydrochloride))
Drug: Topotecan Hydrochloride — Given IV
  Other Names: Evotopin; Hycamptamine; Hycamtin; Nogitecan Hydrochloride; Potactasol; SKF S 104864 A; SKF S-104864-A; SKF S104864A; Topotec; Topotecan HCl; topotecan hydrochloride (oral)
  Arms: Arm I (paclitaxel, doxorubicin, topotecan hydrochloride))

SUMMARY:
This phase II trial studies the possible benefits of treatment with different combinations of the drugs durvalumab, olaparib and cediranib vs. the usual treatment in patients with ovarian, primary peritoneal, or fallopian tube cancer that has come back after a period of improvement with platinum therapy (recurrent platinum resistant). Usual treatment is the type of treatment most patients with this condition receive if they are not part of a clinical study. Combination therapies studied in this trial include MEDI4736 (durvalumab) plus olaparib and cediranib, durvalumab and cediranib, or olaparib and cediranib. Monoclonal antibodies, such as durvalumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumors cells to grow and spread. Olaparib is an inhibitor of PARP, an enzyme that helps repair deoxyribonucleic acid (DNA) when it becomes damaged. Blocking PARP may help keep cancer cells from repairing their damaged DNA, causing them to die. PARP inhibitors are a type of targeted therapy. Cediranib may stop the growth of tumor cells by blocking VEGF (an enzyme). needed for cell growth. Giving different combinations of durvalumab, olaparib and cediranib may work better in increasing the duration of time that the cancer does not progress compared to the usual treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the efficacy of the combinations durvalumab (MEDI4736) plus olaparib and cediranib, durvalumab (MEDI4736) plus cediranib, or olaparib and cediranib, as measured by progression-free survival (PFS), as compared to physician's choice standard of care chemotherapy, in patients with recurrent platinum-resistant ovarian, primary peritoneal or fallopian tube cancer who had prior bevacizumab.

SECONDARY OBJECTIVES:

I. To assess the efficacy of the combinations durvalumab (MEDI4736) plus olaparib and cediranib, durvalumab (MEDI4736) plus cediranib, or olaparib and cediranib, as measured by overall response rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, as compared to physician's choice standard of care chemotherapy, in patients with recurrent platinum-resistant ovarian, primary peritoneal or fallopian tube cancer who had prior bevacizumab.

II. To assess the efficacy of the combinations durvalumab (MEDI4736) plus olaparib and cediranib, durvalumab (MEDI4736) plus cediranib, or olaparib and cediranib, as measured by overall survival (OS), as compared to physician's choice standard of care chemotherapy, in patients with recurrent platinum-resistant ovarian, primary peritoneal or fallopian tube cancer who had prior bevacizumab.

OUTLINE: Patients are randomized to 1 of 4 arms.

ARM I: Patients receive paclitaxel intravenously (IV) over 60 minutes on days 1, 8, and 15, or pegylated liposomal doxorubicin hydrochloride IV over 60 minutes on day 1, or topotecan hydrochloride IV over 30 minutes on days 1, 8 and 15 or days 1-5 per the discretion of the treating physician. Cycles repeat every 21 or 28 days in the absence of disease progression or unacceptable toxicity. Patients may undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) during screening and as clinically indicated on study. Patients also undergo collection of blood and computed tomography (CT) with contrast during screening, and CT or magnetic resonance imaging (MRI) scans throughout the trial.

ARM II: Patients receive durvalumab IV over 60 minutes on day 1, cediranib maleate orally (PO) once daily (QD) Monday through Friday, and olaparib PO twice daily (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients may undergo ECHO or MUGA during screening and as clinically indicated on study. Patients also undergo collection of blood and CT with contrast during screening, and CT or MRI scans throughout the trial.

ARM III: Patients receive durvalumab IV over 60 minutes on day 1 and cediranib maleate PO QD Monday through Friday. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients may undergo ECHO or MUGA during screening and as clinically indicated on study. Patients also undergo collection of blood and CT with contrast during screening, and CT or MRI scans throughout the trial.

ARM IV: Patients receive cediranib maleate PO QD on days 1-28 and olaparib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients may undergo ECHO or MUGA during screening and as clinically indicated on study. Patients also undergo collection of blood and CT with contrast during screening, and CT or MRI scans throughout the trial.

After completion of study treatment, patients are followed up periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Women with recurrent/persistent platinum-resistant ovarian, primary peritoneal, or fallopian tube cancers; platinum-resistant disease is defined as progression within < 6 months from completion of platinum based therapy. The date should be calculated from the last administered dose of platinum therapy
* Patients must have histologically or cytologically confirmed ovarian cancer, peritoneal cancer or fallopian tube cancer and must have a histological diagnosis of high grade serous, grade 3 endometrioid or clear cell carcinoma based on local histopathological findings. Patients with low grade serous, grade 1 or 2 endometrioid, mixed epithelial, undifferentiated carcinoma, or mucinous carcinoma histologies are also eligible, provided that the patient has a known deleterious BRCA1 or BRCA2 mutation identified through testing at a clinical laboratory. Histologic confirmation of the original primary tumor is required via the pathology report (upload of report required). Confirmation of BRCA1 and BRCA2 germline and/or somatic mutation status and hormone receptor (HR) status is required for all entered patients (if available) via testing report (upload of report[s] required)
* Evaluable disease - defined as RECIST 1.1 measurable disease OR non-measurable disease (defined as solid and/or cystic abnormalities on radiographic imaging that do not meet RECIST 1.1 definitions for target lesions OR ascites and/or pleural effusion that has been pathologically demonstrated to be disease-related in the setting of a CA125 >= 2 x upper limit of normal [ULN])
* Prior therapy:

  * At least two prior treatment regimens (including primary therapy) but up to 5 lines of systemic anticancer therapy. Hormonal therapy (such as tamoxifen, aromatase inhibitors) will not count as a previous treatment regimen.
  * Prior use of bevacizumab in the upfront or recurrent setting is required.
  * Prior use of PARP inhibitor is allowed.
  * Prior use of immune checkpoint blockade (e.g., a PD-L1/PD-1inhibitor or a CTLA-4 inhibitor) is allowed
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Hemoglobin > 10 g/dL
* Platelets >= 100,000/mcL
* Creatinine clearance (CrCL) or estimated glomerular filtration rate (eGFR) of > 50 mL/min estimated using either the Cockcroft-Gault equation, the Modification of Diet in Renal Disease Study, or as reported in the comprehensive metabolic panel/basic metabolic panel (eGFR)
* Urine protein: creatinine ratio (UPC) of =< 1
* Total serum bilirubin level =< 1.5 x ULN (patients with known Gilbert's disease who have bilirubin level =< 3 x ULN may be enrolled)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x ULN
* Age >= 18 years
* Body weight > 30 kg
* Adequately controlled blood pressure (systolic blood pressure [SBP] =< 140; diastolic blood pressure [DBP] =< 90 mmHg) on a maximum of three antihypertensive medications. Patients must have a BP of =< 140/90 mmHg taken in the clinic setting by a medical professional within 2 weeks prior to study registration. It is strongly recommended that patients who are on three antihypertensive medications be followed by a cardiologist or a primary care physician for management of BP while on protocol. Patients must be willing and able to check and record daily blood pressure readings. BP cuffs will be provided to patients randomized to the cediranib-containing arms
* Adequately controlled thyroid dysfunction with no symptoms of thyroid dysfunction and normal thyroid stimulating hormone (TSH). If TSH is not within normal range despite no symptoms of thyroid dysfunction, normal free T4 level is required
* Able to swallow and retain oral medications and no gastrointestinal (GI) illnesses that would preclude absorption of olaparib and cediranib as judged by treating physician
* Toxicities of prior therapy (excepting alopecia and vitiligo), should be resolved to less than or equal to grade 1 as per Common Terminology Criteria for Adverse Events (CTCAE) v5.0
* Women of childbearing potential (WOCBP) must agree to use two forms of birth control (hormonal or barrier method of birth control; abstinence). Note: Definition of women of no longer having childbearing potential: Postmenopausal or evidence of non-childbearing status for women of childbearing potential as confirmed by a negative urine or serum pregnancy test within 7 days prior to start of study treatment. Postmenopausal is defined as: Age >= 60 years, or age < 60 with any one or more of the conditions below:

  * Amenorrhoeic for >= 1 year in the absence of chemotherapy and/or hormonal treatments,
  * Luteinizing hormone and/or follicle stimulating hormone and/or estradiol levels in the post-menopausal range,
  * Radiation-induced oophorectomy with last menses > 1 year ago,
  * Chemotherapy-induced menopause with > 1 year interval since last menses,
  * Surgical sterilization (bilateral oophorectomy or hysterectomy)
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry and authorization permitting release of personal health information

Exclusion Criteria:

* Primary platinum-refractory disease defined as progression during first-line platinum-based chemotherapy
* Rising CA-125 only without RECIST 1.1 evaluable disease
* Prior therapy:

  * Patients who have had chemotherapy, investigational drugs or radiotherapy within 3 weeks prior to study registration or those who have not recovered from adverse events due to agents administered more than 3 weeks earlier.
  * Patients may not have had hormonal therapy within 2 weeks of study registration. Patients receiving raloxifene for bone health as per Food and Drug Administration (FDA) indication may remain on raloxifene absent other drug interactions.
  * Prior use of concurrent olaparib and cediranib combination.
  * Patients who have experienced immune-mediated adverse events requiring dose modification or discontinuation.
  * For patients who have received prior PARP inhibitor:

    * Patients who have required dose modification or dose reduction of olaparib will not be eligible, as they will not be able to start this study at full dose.
    * Patients who have required dose reduction of non-olaparib PARP inhibitors for hematologic adverse events will not be eligible (Note: niraparib that is initiated at 200mg daily per weight and platelet guidelines is not considered a dose reduction).
    * Patients who required dose-reduction of non-olaparib PARP inhibitors for non-hematologic adverse events may be eligible after discussion with the Study Chair if the treating investigator feels that they could appropriately receive olaparib at full dose.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 3 months prior to study registration
* Current signs and/or symptoms of bowel obstruction or signs and/or symptoms of bowel obstruction within 3 months of study registration except temporary (< 24 hr) improved with medical management, within last 3 months
* Any prior grade >= 3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE > grade 1
* Dependency on IV hydration or total parenteral nutrition (TPN)
* Pregnant women. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with these drugs, breastfeeding should be discontinued. These potential risks may also apply to other agents used in this study
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with untreated brain metastases, spinal cord compression, or evidence of symptomatic brain metastases or leptomeningeal disease as noted on computed tomography (CT) or magnetic resonance imaging (MRI) scans should not be included on this study, since neurologic dysfunction may confound the evaluation of neurologic and other adverse events. Patients with treated brain metastases and resolution of any associated symptoms must demonstrate stable post-therapeutic imaging for at least 6 months following therapy prior to starting study registration
* Patients who have the following clinical conditions are considered to be at increased risk for cardiac toxicities. Patients with any cardiac history of the following conditions:

  * History of myocardial infarction or myocarditis within six months of study registration
  * Unstable angina
  * Resting electrocardiogram (ECG) with clinically significant abnormal findings.
  * New York Heart Association functional classification of III or IV
* If cardiac function assessment is clinically indicated or performed: left ventricular ejection fraction (LVEF) less than normal per institutional guidelines, or < 55%, if threshold for normal not otherwise specified by institutional guidelines. Patients with the following risk factors should have a baseline cardiac function assessment:

  * Prior treatment with anthracyclines
  * Prior treatment with trastuzumab or T-DM1
  * Prior central thoracic radiation therapy (RT), including RT to the heart
  * History of myocardial infarction within 6 to 12 months (Patients with history of myocardial infarction within 6 months are excluded from the study)
  * Prior history of impaired cardiac function
* History of stroke or transient ischemic attack within six months of study registration
* Clinically significant peripheral vascular disease or vascular disease (aortic aneurysm or aortic dissection)
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of study treatment. Patients must have recovered from any effects of any major surgery and surgical wound should have healed prior to starting treatment. Note: Local surgery of isolated lesions for palliative intent is acceptable
* Evidence of coagulopathy or bleeding diathesis. Therapeutic anticoagulation for prior thromboembolic events, including warfarin, is permitted. Patients receiving warfarin are recommended to have careful monitoring of international normalized ratio (INR)
* Evidence suggestive of myelodysplastic syndrome (MDS) or acute myelogenous leukemia (AML) on peripheral blood smear or bone marrow biopsy, if clinically indicated. No prior allogeneic bone marrow transplant or double umbilical cord blood transplantation (dUBCT)
* Human immunodeficiency virus (HIV) positive patients due to potential drug and drug interactions
* Patients may not use any complementary or alternative medicines including natural herbal products or folk remedies as they may interfere with the effectiveness of the study treatments
* Receipt of live attenuated vaccine within 30 days prior to the first dose of study treatment. Note: Patients, if enrolled, should not receive live vaccine whilst receiving study treatment and up to 30 days after the last dose of study treatment
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (other than atrial fibrillation with controlled ventricular rate), or psychiatric illness/social situations that would limit compliance with study requirements, substantially increase risk of incurring adverse events or compromise the ability of the patient to given written informed consent
* Patients receiving any medications or substances that are strong inhibitors or inducers of CYP3A4. Dihydropyridine calcium-channel blockers are permitted for management of hypertension
* Current or prior use of immunosuppressive medication within 14 days of study registration. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to durvalumab, olaparib, or cediranib
* Patients with active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis [TB] testing in line with local practice), hepatitis B (known positive hepatitis B virus [HBV] surface antigen (HBsAg) result), or hepatitis C. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for hepatitis C virus (HCV) ribonucleic acid (RNA)
* Patients who have a history of (non-infectious) pneumonitis that required steroids, or current pneumonitis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2026-06-14 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jung-min Lee, Principal Investigator — NRG Oncology
Locations (393):
- United States (386):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - John Muir Medical Center-Concord, Concord, California
  - Sutter Davis Hospital, Davis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - City of Hope Antelope Valley, Lancaster, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - City of Hope South Pasadena, South Pasadena, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - City of Hope Upland, Upland, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Sacred Heart Hospital, Pensacola, Florida
  - Northside Hospital, Atlanta, Georgia
  - CTCA at Southeastern Regional Medical Center, Newnan, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Our Lady of the Lake Medical Oncology, Baton Rouge, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Northwell Health Imbert Cancer Center, Bay Shore, New York
  - Island Gynecologic Oncology, Brightwaters, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Summa Health System - Akron Campus, Akron, Ohio
  - Aultman Alliance Community Hospital, Alliance, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Central Ohio Breast and Endocrine Surgery, Gahanna, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - UPMC Hillman Cancer Center at Butler Health System, Butler, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Bristol Regional Medical Center, Bristol, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Thompson Cancer Survival Center - West, Knoxville, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - Houston Methodist West Hospital, Houston, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Houston Methodist The Woodlands Hospital, The Woodlands, Texas
  - Ballad Health Cancer Care - Bristol, Bristol, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Puerto Rico (7):
  - Cancer Center-Metro Medical Center Bayamon, Bayamón
  - HIMA San Pablo Oncologic Hospital, Caguas
  - Doctors Cancer Center, Manatí
  - Instituto Oncologia Moderna Ponce, Ponce
  - San Juan Community Oncology Group, San Juan
  - Centro Comprensivo de Cancer de UPR, San Juan
  - San Juan City Hospital, San Juan

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Paclitaxel, Doxorubicin, Topotecan Hydrochloride)): Patients receive paclitaxel IV over 60 minutes on days 1, 8, and 15, or pegylated liposomal doxorubicin hydrochloride IV over 60 minutes on day 1, or topotecan hydrochloride IV over 30 minutes on days 1, 8 and 15 or days 1-5 per the discretion of the treating physician. Cycles repeat every 21 or 28 days in the absence of disease progression or unacceptable toxicity. Patients may undergo ECHO or MUGA during screening and as clinically indicated on study. Patients also undergo collection of blood and CT with contrast during screening, and CT or MRI scans throughout the trial.
  Biospecimen Collection: Undergo collection of blood
  Computed Tomography: Undergo CT
  Computed Tomography with Contrast: Undergo CT with contrast
  Echocardiography: Undergo ECHO
  Magnetic Resonance Imaging: Undergo MRI
  Multigated Acquisition Scan: Undergo MUGA
  Paclitaxel: Given IV
  Pegylated Liposomal Doxorubicin Hydrochloride: Given IV
  Topotecan Hydrochloride: Given IV
- Arm II (Durvalumab, Cediranib Maleate, Olaparib): Patients receive durvalumab IV over 60 minutes on day 1, cediranib maleate PO QD Monday through Friday, and olaparib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients may undergo ECHO or MUGA during screening and as clinically indicated on study. Patients also undergo collection of blood and CT with contrast during screening, and CT or MRI scans throughout the trial.
  Biospecimen Collection: Undergo collection of blood
  Cediranib Maleate: Given PO
  Computed Tomography: Undergo CT
  Computed Tomography with Contrast: Undergo CT with contrast
  Durvalumab: Given IV
  Echocardiography: Undergo ECHO
  Magnetic Resonance Imaging: Undergo MRI
  Multigated Acquisition Scan: Undergo MUGA
  Olaparib: Given PO
- Arm III (Durvalumab, Cediranib Maleate): Patients receive durvalumab IV over 60 minutes on day 1 and cediranib maleate PO QD Monday through Friday. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients may undergo ECHO or MUGA during screening and as clinically indicated on study. Patients also undergo collection of blood and CT with contrast during screening, and CT or MRI scans throughout the trial.
  Biospecimen Collection: Undergo collection of blood
  Cediranib Maleate: Given PO
  Computed Tomography: Undergo CT
  Computed Tomography with Contrast: Undergo CT with contrast
  Durvalumab: Given IV
  Echocardiography: Undergo ECHO
  Magnetic Resonance Imaging: Undergo MRI
  Multigated Acquisition Scan: Undergo MUGA
- Arm IV (Cediranib Maleate, Olaparib): Patients receive cediranib maleate PO QD on days 1-28 and olaparib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients may undergo ECHO or MUGA during screening and as clinically indicated on study. Patients also undergo collection of blood and CT with contrast during screening, and CT or MRI scans throughout the trial.
  Biospecimen Collection: Undergo collection of blood
  Cediranib Maleate: Given PO
  Computed Tomography: Undergo CT
  Computed Tomography with Contrast: Undergo CT with contrast
  Echocardiography: Undergo ECHO
  Magnetic Resonance Imaging: Undergo MRI
  Olaparib: Given PO
Period: Overall Study
Arm/Group | Arm I (Paclitaxel, Doxorubicin, Topotecan Hydrochloride)) | Arm II (Durvalumab, Cediranib Maleate, Olaparib) | Arm III (Durvalumab, Cediranib Maleate) | Arm IV (Cediranib Maleate, Olaparib)
Started | 18 | 33 | 34 | 35
Completed | 6 | 17 | 11 | 13
Not Completed | 12 | 16 | 23 | 22
Not completed — Adverse Event | 2 | 1 | 4 | 5
Not completed — Never Treated | 2 | 0 | 1 | 1
Not completed — On Treatment | 5 | 9 | 9 | 9
Not completed — Symptomatic Deterioration | 1 | 1 | 3 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 3
Not completed — Other Reason | 1 | 3 | 5 | 4

BASELINE CHARACTERISTICS:
Population: Enrolled Patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Paclitaxel, Doxorubicin, Topotecan Hydrochloride)) | Arm II (Durvalumab, Cediranib Maleate, Olaparib) | Arm III (Durvalumab, Cediranib Maleate) | Arm IV (Cediranib Maleate, Olaparib) | Total
Number analyzed (Participants) | 18 | 33 | 34 | 35 | 120
Age, Customized [Count of Participants; unit: Participants]
  20 - 29 | 0 | 0 | 0 | 0 | 0
  30 - 39 | 0 | 0 | 1 | 1 | 2
  40 - 49 | 0 | 1 | 1 | 3 | 5
  50 - 59 | 5 | 12 | 7 | 7 | 31
  60 - 69 | 9 | 17 | 13 | 18 | 57
  70 - 79 | 4 | 3 | 10 | 6 | 23
  >= 80 | 0 | 0 | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 33 | 34 | 35 | 120
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 1 | 1 | 5
  Not Hispanic or Latino | 18 | 29 | 33 | 33 | 113
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 1 | 1 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2 | 4
  White | 16 | 28 | 30 | 32 | 106
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 1 | 1 | 6
Prior Parp Inhibitor Treatment (Stratification Factor) [Count of Participants; unit: Participants]
  Yes | 9 | 16 | 16 | 18 | 59
  No | 9 | 17 | 18 | 17 | 61
Prior Immune Therapy Treatment (Stratification Factor) [Count of Participants; unit: Participants]
  Yes | 3 | 3 | 2 | 5 | 13
  No | 15 | 30 | 32 | 30 | 107

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: The relationship of randomized treatment assignment to progression free survival. The RECIST 1.1 criteria are used for disease progression. Progression is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: From start of treatment to time of progression or death, whichever occurs first. Median follow-up time was 4.8 months (Inter-Quartile Range: 2.0-7.9 months).
Population: All Randomized Subjects
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Paclitaxel, Doxorubicin, Topotecan Hydrochloride)) | Arm II (Durvalumab, Cediranib Maleate, Olaparib) | Arm III (Durvalumab, Cediranib Maleate) | Arm IV (Cediranib Maleate, Olaparib)
Number analyzed (Participants) | 18 | 33 | 34 | 35
Months | 4.2 [1.9 to 5.0] | 2.6 [2.0 to 4.2] | 2.3 [2.0 to 4.6] | 2.3 [2.1 to 3.9]
Statistical Analysis 1: Comparison: Arm I (Paclitaxel, Doxorubicin, Topotecan Hydrochloride)) vs Arm II (Durvalumab, Cediranib Maleate, Olaparib); Test type: Equivalence — This is the Hazard Ratio of Group 2 compared to Group 1; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.44 to 2.31] — This is the Hazard Ratio of Group 2 compared to Group 1
Statistical Analysis 2: Comparison: Arm I (Paclitaxel, Doxorubicin, Topotecan Hydrochloride)) vs Arm III (Durvalumab, Cediranib Maleate); Test type: Equivalence — This is the Hazard Ratio of Group 3 compared to Group 1; Hazard Ratio (HR) = 1.21, 95% CI 2-sided [0.52 to 2.84] — This is the Hazard Ratio of Group 3 compared to Group 1
Statistical Analysis 3: Comparison: Arm I (Paclitaxel, Doxorubicin, Topotecan Hydrochloride)) vs Arm IV (Cediranib Maleate, Olaparib); Test type: Equivalence — This is the Hazard Ratio of Group 4 compared to Group 1; Hazard Ratio (HR) = 1.34, 95% CI 2-sided [0.58 to 3.08]; This is the Hazard Ratio of Group 4 compared to Group 1

2. Secondary Outcome: Objective Response Rate
Description: Determination of response should take into consideration all target and non-target lesions. Here are the definitions of CR, PR, PD and SD: Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters (i.e. the nadir) while on study. The CI is the Jeffreys interval.
Time Frame: From the start of the treatment until disease progression/recurrence, or termination by the DMC. The median followup time was 4.3 months. The maximum followup time was 11 months. Patients are no longer being assessed.
Population: Patients with measurable disease, a baseline tumor assessment, and at least one on-treatment tumor assessment. The study was terminated for futility of all the experimental arms. Many patients withdrew from treatment prior to their first on-treatment tumor assessment.
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | Arm I (Paclitaxel, Doxorubicin, Topotecan Hydrochloride)) | Arm II (Durvalumab, Cediranib Maleate, Olaparib) | Arm III (Durvalumab, Cediranib Maleate) | Arm IV (Cediranib Maleate, Olaparib)
Number analyzed (Participants) | 10 | 21 | 20 | 18
Proportion of Participants | 0 [0 to 0.217] | 0.048 [0.005 to 0.202] | 0.150 [0.044 to 0.349] | 0.111 [0.024 to 0.311]

3. Secondary Outcome: Duration of Response
Description: Tumor response was assessed using Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1) criteria. Duration of response was defined as the time from the first documentation of objective tumor response (complete response (CR) or partial response (PR)) to the first documented progressive disease (PD), or to death due to any cause, whichever occurs first.
  Per RECIST, Complete Response (CR) is defined as the disappearance of all target lesions; Partial Response (PR) is defined as an >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
  Reporting the number of months from complete or partial response until disease progression, death or censoring, whichever occurs first. In the absence of disease progression or death, censoring time is based on date of last CT scan.
Time Frame: Throughout study treatment, up to 10.6 months.
Population: Patients with Complete or Partial Response
Measure: Median (Full Range); unit: days (censored, progressive disease)
Arm/Group | Arm I (Paclitaxel, Doxorubicin, Topotecan Hydrochloride)) | Arm II (Durvalumab, Cediranib Maleate, Olaparib) | Arm III (Durvalumab, Cediranib Maleate) | Arm IV (Cediranib Maleate, Olaparib)
Number analyzed (Participants) | 0 | 1 | 3 | 2
days (censored, progressive disease) |  | 2.3 [2.3 to 2.3] | 4.1 [2.1 to 5.8] | 6.5 [3.4 to 9.7]

4. Secondary Outcome: Overall Survival
Description: Overall survival will be presented by Kaplan Meier methods. Overall Survival (OS) is defined as the duration of time from study entry to date of death from any cause. A subject who has not died will be censored on the date that they were last known to be alive.
Time Frame: Time from study entry to date of death from any cause, or termination by the DMC. The median followup time was 4.3 months. The maximum followup time was 11 months. Patients are no longer being assessed.
Population: All randomized subjects
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Paclitaxel, Doxorubicin, Topotecan Hydrochloride)) | Arm II (Durvalumab, Cediranib Maleate, Olaparib) | Arm III (Durvalumab, Cediranib Maleate) | Arm IV (Cediranib Maleate, Olaparib)
Number analyzed (Participants) | 18 | 33 | 34 | 35
months | 6.4 [4.8 to NA] — Insufficient number of events to estimate parameter. | 4.9 [3.4 to NA] — Insufficient number of events to estimate parameter. | 5.7 [3.1 to NA] — Insufficient number of events to estimate parameter. | 9.4 [3.4 to NA] — Insufficient number of events to estimate parameter.
Statistical Analysis 1: Comparison: Arm I (Paclitaxel, Doxorubicin, Topotecan Hydrochloride)) vs Arm II (Durvalumab, Cediranib Maleate, Olaparib); Test type: Equivalence — This is the Hazard Ratio of Group 2 compared to Group 1; Hazard Ratio (HR) = 1.41, 95% CI 2-sided [0.44 to 4.47] — This is the Hazard Ratio for Group 2 compared to Group 1
Statistical Analysis 2: Comparison: Arm I (Paclitaxel, Doxorubicin, Topotecan Hydrochloride)) vs Arm III (Durvalumab, Cediranib Maleate); Test type: Equivalence — This is the Hazard Ratio of Group 3 compared to Group 1; Hazard Ratio (HR) = 1.30, 95% CI 2-sided [0.40 to 4.19] — This is the Hazard Ratio of Group 3 compared to Group 1
Statistical Analysis 3: Comparison: Arm I (Paclitaxel, Doxorubicin, Topotecan Hydrochloride)) vs Arm IV (Cediranib Maleate, Olaparib); Test type: Equivalence — This is the Hazard Ratio of Group 4 compared to Group 1; Hazard Ratio (HR) = 1.34, 95% CI 2-sided [0.58 to 3.08] — This is the Hazard Ratio of Group 4 compared to Group 1

5. Secondary Outcome: Count of Participants With a Grade 3 (or Higher) Adverse Event
Description: The number of patients (in each reporting group) who experienced a grade 3 (or higher) adverse event
Time Frame: From the start of treatment until disease progression/recurrence or termination by the DMC. The median followup time was 4.3 months. The maximum followup time was 11 months. Patients are no longer being assessed.
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Paclitaxel, Doxorubicin, Topotecan Hydrochloride)) | Arm II (Durvalumab, Cediranib Maleate, Olaparib) | Arm III (Durvalumab, Cediranib Maleate) | Arm IV (Cediranib Maleate, Olaparib)
Number analyzed (Participants) | 14 | 29 | 26 | 29
Participants | 7 | 19 | 14 | 18

ADVERSE EVENTS:
Time Frame: From the start of treatment until disease progression/recurrence or termination by the DMC. The median followup time was 4.3 months. The maximum followup time was 11 months. Patients are no longer being assessed.
Description: Toxicity assessments will be done using NCI Common Terminology Criteria for Adverse Events (CTCAE v.5). Note: the population for all cause mortality is all randomized subjects. The population for adverse event reporting is the safety population (which has less subjects as it is only treated subjects).
Arm/Group | Arm I (Paclitaxel, Doxorubicin, Topotecan Hydrochloride)) | Arm II (Durvalumab, Cediranib Maleate, Olaparib) | Arm III (Durvalumab, Cediranib Maleate) | Arm IV (Cediranib Maleate, Olaparib)
All-Cause Mortality (participants affected / at risk) | 4/18 | 12/33 | 13/34 | 9/35
Serious Adverse Events (participants affected / at risk) | 8/14 | 19/29 | 14/26 | 18/29
Other Adverse Events (participants affected / at risk) | 12/14 | 25/29 | 24/26 | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Paclitaxel, Doxorubicin, Topotecan Hydrochloride)) (N=14) | Arm II (Durvalumab, Cediranib Maleate, Olaparib) (N=29) | Arm III (Durvalumab, Cediranib Maleate) (N=26) | Arm IV (Cediranib Maleate, Olaparib) (N=29)
Anemia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 0 | 1
Heart failure (Cardiac disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2 | 2
Ascites (Gastrointestinal disorders) | 2 | 1 | 0 | 2
Colonic obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colonic perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 2 | 3
Duodenal obstruction (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 2 | 0 | 3
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 3 | 2 | 2
Death NOS (General disorders) | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 1 | 1 | 0
Fatigue (General disorders) | 1 | 1 | 1 | 5
Fever (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 1
Appendicitis perforated (Infections and infestations) | 0 | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Thrush (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 0
Alkaline phosphatase increased (Investigations) | 1 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Creatinine increased (Investigations) | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 4 | 0 | 0 | 1
Platelet count decreased (Investigations) | 2 | 1 | 0 | 1
White blood cell decreased (Investigations) | 2 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
CELLULITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 2 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Mania (Psychiatric disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
GFR DECREASED (Renal and urinary disorders) | 0 | 1 | 0 | 0
Vaginal fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 6 | 5 | 8
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 1 | 2 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Paclitaxel, Doxorubicin, Topotecan Hydrochloride)) (N=14) | Arm II (Durvalumab, Cediranib Maleate, Olaparib) (N=29) | Arm III (Durvalumab, Cediranib Maleate) (N=26) | Arm IV (Cediranib Maleate, Olaparib) (N=29)
Anemia (Blood and lymphatic system disorders) | 6 | 8 | 3 | 11
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
INCREASED HEMATOCRIT (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 1 | 2
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 2 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 2 | 0
Hypothyroidism (Endocrine disorders) | 1 | 2 | 3 | 2
Blurred vision (Eye disorders) | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1
STYE (Eye disorders) | 0 | 1 | 0 | 0
Watering eyes (Eye disorders) | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 4 | 8 | 6 | 5
Ascites (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Bloating (Gastrointestinal disorders) | 2 | 3 | 1 | 5
Constipation (Gastrointestinal disorders) | 4 | 6 | 4 | 4
Diarrhea (Gastrointestinal disorders) | 6 | 12 | 14 | 17
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 2 | 2
Gastroparesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
HEARTBURN (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Ileal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 2 | 4 | 4
Nausea (Gastrointestinal disorders) | 4 | 14 | 6 | 18
Rectal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 8 | 2 | 7
BILATERAL LOWER EXTREMITY EDEMA (General disorders) | 0 | 0 | 0 | 1
CHEST TIGHTNESS (General disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 1 | 2 | 0
Edema limbs (General disorders) | 1 | 3 | 2 | 7
Facial pain (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 5 | 18 | 8 | 13
Fever (General disorders) | 1 | 1 | 2 | 2
Flu like symptoms (General disorders) | 0 | 0 | 1 | 1
GENERALIZED BODY ACHES (General disorders) | 0 | 1 | 0 | 0
Generalized edema (General disorders) | 1 | 0 | 0 | 0
LEFT LOWER EXTREMITY EDEMA (General disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 0 | 1
NUMBNESS AND TINGLING (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 1
Pain (General disorders) | 0 | 1 | 1 | 5
Autoimmune disorder (Immune system disorders) | 0 | 0 | 1 | 0
Bronchial infection (Infections and infestations) | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 2
Eye infection (Infections and infestations) | 0 | 1 | 0 | 0
INFECTION GENERAL (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 2
Skin infection (Infections and infestations) | 0 | 0 | 0 | 2
Thrush (Infections and infestations) | 0 | 1 | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 1 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 2 | 0
BROKEN TOE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 2 | 0
Alkaline phosphatase increased (Investigations) | 3 | 4 | 2 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 3 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1
Cardiac troponin I increased (Investigations) | 1 | 0 | 0 | 0
Creatinine increased (Investigations) | 2 | 9 | 3 | 7
Hemoglobin increased (Investigations) | 0 | 1 | 0 | 0
INR increased (Investigations) | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 3 | 1 | 2 | 2
Neutrophil count decreased (Investigations) | 4 | 2 | 1 | 2
Platelet count decreased (Investigations) | 4 | 4 | 2 | 8
Thyroid stimulating hormone increased (Investigations) | 0 | 4 | 3 | 2
Weight loss (Investigations) | 1 | 3 | 6 | 5
White blood cell decreased (Investigations) | 4 | 5 | 2 | 4
Anorexia (Metabolism and nutrition disorders) | 2 | 10 | 2 | 9
Dehydration (Metabolism and nutrition disorders) | 1 | 3 | 1 | 3
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 3 | 4 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 3 | 2 | 1
Hypokalemia (Metabolism and nutrition disorders) | 3 | 3 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 1 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 3 | 3 | 3 | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2
LOSS OF BALANCE (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 2
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 5 | 3 | 5
Dysgeusia (Nervous system disorders) | 2 | 3 | 3 | 3
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 6 | 6 | 9
Memory impairment (Nervous system disorders) | 0 | 0 | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 4
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 3
Confusion (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 2
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 1 | 0 | 1
GFR DECREASED (Renal and urinary disorders) | 0 | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 1 | 0 | 1
LOW URINE OUTPUT (Renal and urinary disorders) | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 2 | 1 | 4
Urinary frequency (Renal and urinary disorders) | 0 | 1 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 2
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 2 | 0 | 0
Vaginal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 6 | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 6 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 3 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
EXCORIATION OF PERINEAL AREA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
FACIAL PIMPLES (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Nail changes (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 6 | 1 | 1
SKIN PEELING- BILATERAL FEET (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
DEEP VEIN THROMBOSIS RIGHT LOWER EXTREMITY (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 3 | 13 | 9 | 14
Hypotension (Vascular disorders) | 1 | 0 | 1 | 2
Thromboembolic event (Vascular disorders) | 0 | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT04739800/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-23): https://cdn.clinicaltrials.gov/large-docs/00/NCT04739800/ICF_001.pdf